CLINICAL TRIAL: NCT01303003
Title: Evaluation of Addition of Dexamethasone to Transversus Abdominis Plane (TAP) Peripheral Nerve Block: Does it Enhance the Quality and Duration of Analgesia?
Brief Title: Evaluation of Addition of Dexamethasone to Transversus Abdominis Plane (TAP) Peripheral Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TAP-00560
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Prostate CA
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm 1 (Experimental): Bilateral TAP block consisting of 40cc. 0.125% bupivicaine + 0.5cc. dexamethasone (2mg.) per side.
  Interventions: Drug: Dexamethasone
- Treatment Arm 2 (Active Comparator): Bilateral TAP block of 40cc. of 0.125% bupivicaine + 0.5cc. sterile saline per side
  Interventions: Procedure: TAP block

INTERVENTIONS:
Drug: Dexamethasone — 40 cc. 0.125% bupivicaine + 0.5cc. dexamethasone (2mg.) per side.
  Arms: Treatment Arm 1
Procedure: TAP block — Bilateral TAP block of 40cc. of 0.125% bupivicaine + 0.5cc. sterile saline per side
  Arms: Treatment Arm 2

SUMMARY:
Transversus abdominis plane (TAP) blocks are increasingly being performed after abdominal surgery to provide post operative analgesia. Dexamethasone has demonstrated an ability to prolong the effective duration of analgesia in several different peripheral nerve blocks. The study will examine, in a blinded, prospective and randomized fashion, whether the addition of dexamethasone to TAP blocks similarly prolongs blockade and pain relief. The study will compare local anesthetic with and without the addition of dexamethasone in the TAP block.

DETAILED DESCRIPTION:
The study will be done in two phases. In the first phase, patients will be randomized to receive either 20 cc of 0.125% bupivicaine with or without 2 mg of dexamethasone on each side of their abdomen (40 cc and 4 mg in total) and patients who receive the dexamethasone will be compared with patients who did not receive it. In the second phase, we will assess whether patients can serve as their own controls by adding dexamethasone only to one side of the block (one side of the abdomen) and comparing pain relief/efficacy with the contra-lateral plain local anesthetic effect. The study will assess pain relief, opioid consumption, level of blockade, and operator's prospective assessment of likely efficacy, based on the ultrasound visualization of the local anesthetic injection as compared with actual efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients, between ages 18-85 years old, undergoing Robot-assisted laparoscopic prostatectomy by a single surgeon at a single hospital.
* Subjects are physically and mentally able to participate in the study.
* Subjects are able to give fully informed consent to participating in this study after demonstrating good understanding of the risks and benefits of the proposed components of the TAP block.

Exclusion Criteria:

* Demonstrated hypersensitivity or allergy to local anesthetics or dexamethasone.
* Any subject whose anatomy, or surgical procedure, in the opinion of the investigator, might preclude the potential successful performance of a TAP block.
* Any subject, who in the opinion of the investigator, might be harmed or be a poor candidate for participation in the study.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sternlicht, MD, Principal Investigator — St. Elizabeth's Medical Center of Boston
Locations (1):
- St. Elizabeth's Medical Center of Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No data are available for this study, due to the fact that the PI has left the institution. Multiple efforts were made, by Research and senior leadership, to contact the PI, prior to and after his leaving the institution, with no response. Sincere efforts were made to obtain the data for reporting, but the data is unavailable.
Period: Overall Study
Arm/Group | Treatment Arm 1 | Treatment Arm 2
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data are available for this study, due to the fact that the PI has left the institution. Multiple efforts were made, by Research and senior leadership, to contact the PI, prior to and after his leaving the institution, with no response. Sincere efforts were made to obtain the data for reporting, but the data is unavailable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm 1 | Treatment Arm 2 | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Time to First Request of Additional Analgesia
Description: Documenting the time required by patients to the first request of additional analgesia.
Time Frame: 24 hours post-op
Population: as for baseline characteristics
Arm/Group | Treatment Arm 1 | Treatment Arm 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Assess the Efficacy of the TAP Block by Measuring Visual Analog Scales, Total Opioid Use During the First 24 Hours Post-op, and Provider Assessments to Recognize the Overall Efficacy of the Procedure With and Without Dexamethasone Adjunct.
Time Frame: 24 hours post-op
Population: No data are available for this study, due to the fact that the PI and study staff have left the institution. Multiple efforts were made, by Research and senior leadership, to contact the PI, prior to and after his leaving the institution, with no response. Sincere efforts were made to obtain the data for reporting, but the data is unavailable.
Arm/Group | Treatment Arm 1 | Treatment Arm 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No data are available for this study, due to the fact that the PI has left the institution. Multiple efforts were made, by Research and senior leadership, to contact the PI, prior to and after his leaving the institution, with no response. Sincere efforts were made to obtain the data for reporting, but the data is unavailable.
Arm/Group | Treatment Arm 1 | Treatment Arm 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes